CLINICAL TRIAL: NCT03200470
Title: The Utility of Next-generation Sequencing for the Diagnosis of Periprosthetic Joint Infection
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Other Study IDs: 2017JPAR
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Prosthetic Joint Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Suspected PJI
  Interventions: Other: No intervention: sample collection study

INTERVENTIONS:
Other: No intervention: sample collection study — Sample collection and collection of laboratory values

SUMMARY:
This is a prospective multicenter study. All patients presenting for revision hip or knee arthroplasty for all indications under the respective surgeon's care may be eligible. Per standard of care preoperatively, all patients must have blood drawn for erythrocyte sedimentation rate(ESR), C-reactive protein(CRP) and D-dimer. Aspiration of the joint in question may be performed at the discretion of the treating surgeon and results documented. Intraoperative samples will also be collected and sent for NGS analysis

DETAILED DESCRIPTION:
Pre-operative D-dimer testing should be performed if this is in keeping with the local institutional standard of care. Otherwise, D-dimer testing will be omitted from the pre-operative panel of tests collected.

NGS results will be made available to the Investigator. Treatment will remain within keeping with the Investigator's standard of care. NGS results may be used at the discretion of the treating surgeon in guiding patient treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing primary total hip or knee arthroplasty with no history of prior surgery
2. Patients undergoing revision hip or knee arthroplasty for septic or aseptic indication.

Exclusion Criteria:

1. Patients undergoing second stage re-implantation surgery for PJI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Samples will be collected from subjects undergoing revision for suspected infection. Data analysis will occur on samples collected
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-02-16 (Actual); Primary Completion 2018-02 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
NextGeneration Sequencing analysis concordance with Muskuloskeletal Infection Society (MSIS) criteria for defining infection | Immediate post-operative period (usually within 5 days following surgery)
  MSIS criteria incorporates pre-operative laboratory values with tissue and fluid samples collected during surgery in an attempt to diagnose infection

CONTACTS AND LOCATIONS:
Overall Officials: Tiffany Morrison, MS, CCRP, Study Chair — Rothman Institute
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States